CLINICAL TRIAL: NCT00130143
Title: Open-Label Prospective Trial Evaluating the Toxicities Associated With Subcutaneous Administration of Ethyol (Amifostine) for the Prevention of Radiation-Induced Toxicities
Brief Title: Toxicities Associated With Subcutaneous Administration of Ethyol (Amifostine) for the Prevention of Radiation-Induced Toxicities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Dale & Frances Hughes Cancer Center (Other)
Collaborators: MedImmune LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ethyol Study #ETH156-03D
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2005-09-27 (Estimated); Status verified 2005-08

CONDITIONS: Head and Neck Cancer; Lung Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms | interventions — Amifostine

INTERVENTIONS:
Drug: Ethyol (Amifostine)

SUMMARY:
Dry mouth occurs very often in patients who receive radiation treatment. Amifostine is a drug approved to reduce the short and long-term occurrence of dry mouth when patients receive radiation treatment for head and neck cancer. Some studies have shown that Amifostine reduces the side effects of radiation treatment for lung cancer. The use of Amifostine is still being investigated in lung malignancies. Amifostine is found to be a protectant from radiation side effects of such normal tissues as bone marrow, skin, oral mucosal, esophagus, kidney and testes. Patients that receive radiation treatments for lung cancer may experience side effects involving the esophagus. It is hoped that patients will benefit from the protection of their esophagus and avoid delays in radiation treatment due to side effects of the radiation.

DETAILED DESCRIPTION:
The protective capacity of thio-containing compounds against normal tissue damage from radiation have been recognized for over 40 years..

Although intravenous administration is the approved standard route, because of practical advantages there has been increasing interest in the subcutaneous administration of Ethyol, which presents multiple advantages when used for radioprotection.

Based on the data that has been presented, as well as the personal experience of this and other physicians/centers with subcutaneous administration of amifostine, the researchers are proposing an open-label study evaluating the rate and severity of toxicities associated with this route of administration. Toxicities to be assessed include nausea/vomiting, hypotension, and skin/fever reactions.

ELIGIBILITY:
Inclusion Criteria:

* Patient is eligible to receive subcutaneous amifostine under site's current practice guidelines for radioprotection.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Age > 18
* Patient receiving radiation therapy or combined modality therapy to treat malignancy.
* No evidence of distant metastatic disease.
* Granulocyte count (segs & bands) > 2000/mm3 and platelet count > 100,000/mm3
* Serum creatinine <2.0mg/dL
* Total bilirubin <2.0mg%, SGOT < times the upper limit of normal.
* Patients may not be entered on investigational therapeutic trials.
* Patients or guardians must be informed of and understand the investigational nature of this study and give written informed consent prior to any study procedures.

Exclusion Criteria:

* Life expectancy of <6 months
* Patients receiving only chemotherapy to treat malignancy.
* Patients who have been treated with any investigational drugs <4 weeks prior to study entry.
* General medical or psychological conditions which would not permit the patient to complete the study or sign the informed consent.
* Pregnancy; Women of childbearing potential should use an effective (for them) method of birth control throughout their participation in this study.
* Patients who are currently receiving or have received amifostine for radioprotection within the prior 6 months are excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-06; Study Completion 2004-09

PRIMARY OUTCOMES:
Primary endpoint: To evaluate how amifostine is given subcutaneously at each institution
To determine treatment related toxicities and safety of subcutaneous administration of amifostine for the prevention of radiation-induced toxicities

SECONDARY OUTCOMES:
Secondary endpoints: Evaluate efficacy of amifostine in reducing radiation induced toxicities in these patients

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Greenberg, M.D., Principal Investigator — The Dale & Frances Hughes Cancer Center
Locations (1):
- The Dale & Frances Hughes Cancer Center, East Stroudsburg, Pennsylvania, United States